CLINICAL TRIAL: NCT00372710
Title: Efficacy and Tolerability of Intravenous Zoledronic Acid 4mg as an Adjunct to Standard Therapies Including Conversion From Pamidronate in Breast Cancer Patients With Metastatic Bone Lesions. A Prospective, Randomised, Open-label, Clinical Study
Brief Title: Safety/Efficacy of Intravenous Zoledronic Acid When Added to Standard Therapies in Patients With Breast Cancer and Metastatic Bone Lesions
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CZOL446EDE03
Record Dates: First submitted 2006-09-06; First posted 2006-09-07 (Estimated); Last update posted 2009-11-23 (Estimated); Status verified 2009-11

CONDITIONS: Breast Cancer With Bone Metastasis
Keywords: Breast cancer; Palliation; Bone metastasis; Zoledronic acid
MeSH Terms: conditions — Breast Neoplasms | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic acid

SUMMARY:
Zoledronic acid selectively binds to bone and protects it from being metastasized by tumor cells. This study evaluates the safety and efficacy of zoledronic acid when added to standard therapies in breast cancer patients with metastatic bone lesions.

ELIGIBILITY:
Inclusion criteria

* Confirmed diagnosis of Breast Cancer with at least one breast cancer-related bone lesion
* No treatment with bisphosphonates within 6 months prior to inclusion into the study
* Good health status (ECOG Performance status 0-2)

Exclusion criteria

* Patients who do not have at least one breast cancer-related bone lesion that is detectable on conventional radiographs of bone (plain film) at screening
* Abnormal renal function
* History of diseases with influence on bone metabolism such as Paget's disease and primary hyperparathyroidism
* Pregnancy and lactation
* Current active dental problems including infection of the teeth or jawbone (maxilla or mandibular); dental or fixture trauma, or a current or prior diagnosis of osteonecrosis of the jaw (ONJ), of exposed bone in the mouth, or of slow healing after dental procedures, recent (within 6 weeks) or planned dental or jaw surgery (e.g..extraction, implants)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2002-08

PRIMARY OUTCOMES:
Efficacy of a switch over from pamidronate therapy (2 infusions) to a treatment with zoledronic acid 4mg every 4 weeks (10 infusions) for 44 weeks in patients with breast cancer-related bone lesions

SECONDARY OUTCOMES:
Comparison of the safety, tolerability, and efficacy in the treatment arms

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Chair — Novartis
Locations (1):
- Freiburg im Breisgau, Germany